CLINICAL TRIAL: NCT03047499
Title: Evaluation of the Effect of Botulinum Toxin Type-A Injection Prior to Surgical Correction of Complete Unilateral Cleftlip Repair by Modified Millard Cheiloplasty
Brief Title: Evaluation of the Effect of Botulinum Toxin Type-A Injection Prior to Surgical Correction of Complete Unilateral Cleft Lip Repair by Modified Millard Cheiloplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mostafa Khairy (Other)
Responsible Party: Sponsor-Investigator, Mostafa Khairy, Mostafa Khairy, Cairo University
Organization: Cairo University (Other)
Other Study IDs: CEBC-CU-2017-02-04
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Esthetic Outcome of Injection of Botulinum Toxin Type-A in Cleft Lip Repair
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Scar Length
  Interventions: Drug: Botulinum toxin type A
- Vancouver scar scale
  Interventions: Drug: Botulinum toxin type A
- Scar width
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — Botulinum toxin type-A injection

SUMMARY:
Evaluation of the effect of botulinum toxin type-A injection prior to surgical correction of complete unilateral cleftlip repair by modified millard cheiloplasty

ELIGIBILITY:
Inclusion Criteria:

* Primary cleft lip

Exclusion Criteria:

* Cleft palate

Ages: 3 Months to 6 Months | Sex: All
Age Groups: Child
Study Population: Children up to 6 months
Sampling Method: Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2017-02-15 (Estimated); Primary Completion 2017-10-15 (Estimated); Study Completion 2017-11-15 (Estimated)

PRIMARY OUTCOMES:
Scar Length | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt